CLINICAL TRIAL: NCT00792506
Title: Phase II High Pulse Dose Clinical Trial of Orally Administered ITF2357 In Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Phase II Clinical Trial of ITF2357 In Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely discontinued for lack of recruitement.
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DSC/07/2357/29; 2008-001416-20 (EudraCT Number)
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — givinostat hydrochloride; Histone Deacetylase Inhibitors

STUDY DESIGN:
Masking Description: This was an open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- ITF2357 (Experimental): Eligible patients had to be treated with weekly single doses of ITF2357 according to the above mentioned treatment plan.
  Interventions: Drug: ITF2357

INTERVENTIONS:
Drug: ITF2357 — Treatment was to be administered on an inpatient basis from week 1 to week 13 and on an outpatient basis from week 14 to anticipated end of treatment (week 18). The patients had to be hospitalized on day 1 every week. The Investigator had to administer ITF 2357 in one single dose (two or three 200 mg capsules at one time) under his/her direct control.
  Other Names: Histone-Deacetylase Inhibitor

SUMMARY:
Primary objective:

To assess the safety of ITF 2357 administered once weekly at high pulse dose in patients with relapsing/refractory multiple myeloma.

Secondary objectives:

1. To evaluate the anti-tumour activity of ITF 2357 administered once weekly at high pulse dose in patients with advanced multiple myeloma, measured as decrease of M protein.
2. To assess the therapeutic response to ITF3257 according to EBMT criteria.
3. To determine pharmacokinetic profile of ITF 2357 administered following high pulse dose schedule.

DETAILED DESCRIPTION:
This is open label, phase IIa High Pulse Dose Clinical Trial testing ITF2357 (orally administered) in adult patients with relapsing/refractory multiple myeloma after at least 2 previous lines of treatment.

Patients are planned to receive ITF2357 in accordance with following scheme:

Weeks 1-6

Patient #01 is planned to receive ITF 2357 at 400 mg in one single dose on day 1, 8, 15, 22, 29 and 36. Safety assessments are planned to be performed twice a week. If no issue (grade >3 neutropenia or any other grade ≥3 toxicity) emerges at day 15, two further patients (#02 and #03) will be enrolled and receive the same dose. If patients #02 and #03 show a favourable safety profile at day 15, and in the meantime no safety concerns arise from patient #01, the further patients will be enrolled and treated according to the below reported scheme:

* 8 more patients (#04-11) will receive 400 mg once weekly; safety assessments will be performed weekly.
* 1 patient (#12) will receive 600 mg once weekly; safety assessments will be performed twice a week.

If no safety concern emerges from patient 12 at day 15, two further patients (#13 and #14) will be enrolled and treated with 600 mg once weekly. If patients #13 and #14 don't show relevant safety concerns (grade >3 neutropenia or any other grade ≥3 toxicity) at day 15, and in the meanwhile patient #12 maintains a favourable safety profile, eight further patients (#15-22) will be recruited and receive the same treatment regimen.

If grade >3 neutropenia or any other grade ≥3 toxicity appear at any time during week 1-6, the treatment will be permanently discontinued.

In this phase, treatment will be administered on an inpatient basis.

Weeks 7-12

For patients still on therapy at day 43 visit, M protein will be quantified and the treatment continued or possibly modified as follows on the basis of this parameter:

Decrease >or= of 25%:

patients in 400/week group continue 400mg for 6 further weeks patients in 600/week group continue 600mg for 6 further weeks

Stable +or- of 25%:

patients in 400/week group increase to 600mg and continue for 6 further weeks patients in 600/week group add dexamethasone 40mg for 4 days/week (day 1-4) and continue 600mg for 6 further weeks

Increase > of 25%:

patients in 400/week group add dexamethasone 40mg for 4 days/week (day 1-4) and continue 400mg for 6 further weeks patients in 600/week group failure:out of the study patients in 600/week group

Safety assessments will be performed at weekly intervals. In case of grade >3 neutropenia or any other grade ≥3 toxicity the treatment will be permanently discontinued.

In this phase treatment will be administered on an inpatient basis.

Weeks 13-18

For patients still on therapy at day 85 (week 13, day 1), the response rate will be quantified according to EBMT criteria. In case of response (complete, partial or minimal) or stable disease (no change) the treatment will be prolonged until week 18, whereas in case of disease progression the patient will leave the study. A new complete efficacy evaluation will be performed at day 127 (end of treatment).

During this phase safety will be assessed at weekly intervals and in case of grade >3 neutropenia or any other grade ≥3 toxicity the treatment will be permanently discontinued.

This phase of the study will be conducted on an outpatient basis.

No dosage modification or temporary discontinuation is admitted.

Only one patient has been enrolled. The drug was ineffective in determining an improvement of the patient's disease status according to the EBMT response criteria.The study was prematurely discontinued for lack of recruitment.No firm conclusion on the safety and efficacy of ITF2357 administered at high (400 or 600 mg) single weekly doses can be drawn from the data collected from the only one patient recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of multiple myeloma according to International Myeloma Working Group diagnostic criteria
2. Age ≥ 18 years
3. Patient relapsed after at least 2 lines of conventional chemotherapy or high dose therapy with autologous or allogeneic stem cell support, and/or for whom no alternative treatments are available/suitable
4. Increasing trend of monoclonal immunoglobulin or Bence-Jones proteinuria through the last 4 consecutive pre-screening measurements, already available in the patient history
5. No chemotherapy or other investigational anticancer therapy for at least 3 weeks before the start of the study
6. Full recovery from previous toxicities
7. ECOG performance status 0-2
8. Adequate bone marrow reserve: absolute neutrophil count ≥ 1000/ml; platelet count ≥ 90000/ml
9. Adequate liver function: total bilirubin within normal institutional limits (PI center); AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limit of normal (PI center)
10. Adequate renal function: Creatinine ≤ 2.5 mg/dl or creatinine clearance ≥ 50 ml/min
11. Either men or women, accepting to practice effective contraception during the entire study period unless documentation of infertility exists. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should immediately inform her treating physician; in this case ITF 2357 treatment will be promptly discontinued
12. Able to understand and willing to sign the informed consent form.

Exclusion Criteria:

1. Planned autologous or allogeneic bone marrow transplantation within 4 weeks of the initiation of ITF 2357 administration
2. Concurrent use of medicines that would confound the interpretation of toxicities and anti-tumour activity of ITF 2357 (i.e. quinolones, macrolides, 5-HT3 antagonists except for palonosetron,)
3. Clinically significant illness including, but not limited to, the following: active infection, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, cardiac arrhythmia (present or documented in the past, of any kind), any other condition (including laboratory abnormalities) that in the opinion of the Investigator places the patient to unacceptable risk for adverse outcome if he/she were to participate in the study
4. Psychiatric illness/social situations that would limit compliance with study medication and protocol requirements
5. Pregnant or lactating women
6. Positive blood tests for HIV, HBV, HCV, active EBV and CMV
7. Diseases related to active viral infections
8. Patients with a marked baseline prolongation of QTc interval (e.g. repeated demonstration of a QTc interval >440 ms for men and >450 ms for women)
9. Patients with history of additional risk factors for Torsade de Pointes (e.g. heart failure, family history of Long QT Syndrome).
10. The use of concomitant medications with potential risk of Torsade de Pointes and/or that can prolong QTc interval

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with relapsing/refractory multiple myeloma with TEAE, included serious AE | 30 weeks
  Number of patients with TEAE, included serious AE, was assessed while receiving once weekly ITF2357 at high pulse dose.

SECONDARY OUTCOMES:
Decrease in M protein and clinical response rate (PR plus CR according to the European Group for Blood & Marrow Transplantation - EBMT- criteria). | 18 weeks
  Anti-tumour activity of ITF 2357 was measured as decrease of M protein. While the clinical response rate was represented by a Partial or complete response according to the EBMT criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio La Nasa, MD, Principal Investigator — Presidio Ospedaliero R. Binaghi, Cagliari - Italy
Locations (1):
- Presidio Ospedaliero R. Binaghi, Cagliari, Italy